CLINICAL TRIAL: NCT05608174
Title: Comparison of Tracheal Temperature Measured Using Endotracheal Tube (ETT) Thermometer Before and After Neck Hyperextension in Patients Undergoing Laryngeal Microsurgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0777
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Patients With Laryngeal Microsurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After entering the operating room, the subject receives normal general anesthesia. The operating room temperature should be maintained at 20-25°C, and a blanket is covered and a bare warmer is applied to prevent the patient's body temperature from falling. Check the loss of consciousness due to the administration of intravenous anesthetics, and tracheostomy is performed with a tracheostomy tube (internal diameter: 7.5 mm for male patients and 6.5 mm for female patients) with a temperature measurement sensor embedded in the cuff surface 3 minutes after the administration of muscle relaxant. Immediately after the tracheal tube, air is injected into the cuff of the tracheal tube, and the pressure is 20 cmH2O or less. The depth of the tracheal tube is fixed to 24 cm for male patients and 22 cm for female patients based on teeth. After tracheal intubation, water ventilation is performed, and the end of exhalation carbon dioxide partial pressure (EtCO2) and chest movement are observed to confirm the success of tracheal intubation. Check whether the depth of the tracheal tube is appropriate through auscultation of the lung fields on both sides, and then start machine breathing. Apply a single breath (4-8 ml/kg, expected weight basis) to the mixed gas of oxygen (50%) and air (2L/min), and adjust the number of breaths per minute for EtCO2 40 cmH2O. In order to maintain anesthesia, sevoflurane and repeatanil are administered during surgery. During surgery, SpO2 is maintained at 95% or more, blood pressure and heart rate are maintained at ± 30% of blood pressure and heart rate just before anesthesia, and airway pressure is maintained at 35 cmH2O or less. To compare with the bronchial temperature measured by the bronchial tube thermometer, the esophageal thermometer is inserted to measure the esophageal body temperature. The depth of the esophageal thermometer is determined using the following formula derived from previous studies. Determination of esophageal probe insertion length based on standing and sitting height. (The esophageal thermometer depth (cm) = 0.228 x height - 0.194). Study the temperature measured by the bronchial tube thermometer and the esophageal thermometer. It is the bronchial body temperature measured with a bronchial tube thermometer before and after cervical overstretch. The tracheal body temperature before and after cervical overstretch is defined as the tracheal body temperature just before cervical overstretch and 5 minutes after overstretch, respectively. Record the maximum difference between esophageal and tracheal temperatures before and after cervical hyperplasia, from 5 minutes after bronchial tube thermometer and just before cervical hyperplasia, and from 5 minutes after cervical hyperplasia to end of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The American Anesthesiology Association's Systemic Condition Classification 1, 2, adult patients aged 19 or older, who are scheduled to perform general anesthesia for laryngeal microoperation
2. If the study participant voluntarily decides to participate and agrees in writing after hearing and fully understanding the detailed explanation of this clinical study

Exclusion Criteria:

1. In case the bronchial tube thermometer cannot be used for surgery
2. If you have a history of cervical surgery
3. In the case where neck overstretching for laryngeal microoperation is impossible
4. If the body temperature measured before surgery is 37.6℃ or higher or 35.6℃ or lower
5. Where the researcher determines that it is inappropriate to participate in clinical research due to other reasons;

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who are scheduled to undergo laryngeal micro-surgery under general anesthesia at Yonsei University Severance Hospital.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change of tracheal temperature measured using Endotracheal tube (ETT) thermometer before and after neck hyperextension in patients undergoing laryngeal microsurgery | up to 1 year
  It is the bronchial body temperature measured with a bronchial tube thermometer before and after cervical overstretch. The tracheal body temperature before and after cervical overstretch is defined as the tracheal body temperature just before cervical overstretch and 5 minutes after overstretch, respectively.

SECONDARY OUTCOMES:
The maximum difference between esophageal and bronchial temperatures before and after cervical hyperplasia | up to 1 year
  The maximum difference between esophageal and bronchial temperatures before and after cervical hyperplasia is recorded when esophageal and bronchial temperatures differ the most from 5 minutes after bronchial tube thermometers and just before cervical hyperplasia to end of surgery.

IPD SHARING:
Plan to Share IPD: No